CLINICAL TRIAL: NCT02685345
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, add-on Study of DS-8500a in Japanese Patients With Type 2 Diabetes Mellitus Receiving Sitagliptin
Brief Title: A Study of DS-8500a in Japanese Subjects With Type 2 Diabetes Mellitus Receiving Sitagliptin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Mediscience Planning, Inc. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS8500-A-J204
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; sitagliptin; adult; Phase 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — firuglipel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DS-8500a 25 mg QD (Experimental): DS-8500a 25 mg tablets, orally, once daily (QD) for up to 28 days
  Interventions: Drug: DS-8500a 25 mg
- DS-8500a 75 mg QD (Experimental): DS-8500a 75 mg tablets, orally, once daily (QD) for up to 28 days
  Interventions: Drug: DS-8500a 75 mg
- placebo (Placebo Comparator): placebo tablets, orally, once daily for up to 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-8500a 25 mg
  Arms: DS-8500a 25 mg QD
Drug: DS-8500a 75 mg
  Arms: DS-8500a 75 mg QD
Drug: placebo
  Arms: placebo

SUMMARY:
The objectives of the study is to evaluate the efficacy and safety of DS-8500a compared with placebo in patients with type 2 diabetes mellitus (T2DM) receiving sitagliptin.

DETAILED DESCRIPTION:
In patients with type 2 diabetes mellitus being treated with sitagliptin, efficacy and safety of DS-8500a are to be evaluated after 28-day multiple oral administration of DS-8500a at 25 or 75 mg, in a double-blind, placebo-controlled, parallel-group comparison study.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with type 2 diabetes
* Patients aged ≥ 20 years at the time of informed consent
* Patients who have been treated with sitagliptin 50 mg monotherapy for the treatment of type 2 diabetes mellitus
* Patients who have HbA1c ≥ 7.0% and < 9.0%

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or with a history of diabetic coma, precoma, or ketoacidosis
* Patients receiving or requiring treatment with insulin
* Patients with a body mass index (BMI) of < 18.5 kg/m2 or ≥ 35.0 kg/m2
* Patients with clinically evident renal impairment (estimated glomerular filtration rate [eGFR] of < 45 mL/min per 1.73 m2) or clinically significant renal disease
* Patients with fasting plasma glucose ≥ 240 mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in 24 hour weighted mean glucose | baseline (Day -1) to Day 28

SECONDARY OUTCOMES:
change in fasting plasma glucose | baseline (Day -1) to Day 28
change in plasma glucose | baseline (Day -1) and Day 28
  Day -1 and Day 28: Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast; 0.5, 1, 2, and 4 hours after starting lunch before evening meal; 0.5, 1, 2, and 4 hours after starting evening meal
change in glycoalbumin | baseline (Day -1) and Day 28
change in serum insulin | baseline (Day -1) and Day 28
  Day -1 and Day 28: Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast; 0.5, 1, 2, and 4 hours after starting lunch before evening meal; 0.5, 1, 2, and 4 hours after starting evening meal
change in proinsulin | baseline (Day -1) and Day 28
change in C-peptide | baseline (Day -1) and Day 28
  Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast
change in PYY (pancreatic peptide YY3-36) | baseline (Day -1) and Day 28
  Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast
change in total GLP-1 (Glucagon-like peptide-1) | baseline (Day -1) and Day 28
change in active GLP-1 (Glucagon-like peptide-1) | baseline (Day -1) and Day 28
  Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast
change in total GIP (Gastric inhibitory polypeptide) | baseline (Day -1) and Day 28
  Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast
change in total glucagon | baseline (Day -1) and Day 28
  Before breakfast; 0.5, 1, 2, and 4 hours after starting breakfast
change in total total cholesterol | baseline (Day -1) to after dosing on Day 28
change in total HDL (high density lipoprotein) cholesterol | baseline (Day -1) to after dosing on Day 28
change in total LDL (low density lipoprotein) cholesterol | baseline (Day -1) to after dosing on Day 28
change in total triglyceride | baseline (Day -1) to after dosing on Day 28
number and severity of adverse events | baseline (Day -1) to after dosing on Day 28
change in derived plasma glucose AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from plasma glucose; AUC0-24h, AUC 0-4h, AUC4-8h, AUC9-13h
change in derived serum insulin AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from serum insulin; AUC0-24h, AUC 0-4h, AUC4-8h, AUC9-13h
change in derived C-peptide AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from C-peptide; AUC0-4h
change in derived PYY AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from PYY; AUC0-4h
change in derived total GLP-1 AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from total GLP-1; AUC0-4h
change in derived active GLP-1 AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from active GLP-1; AUC0-4h
change in derived total GIP AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from total GIP; AUC0-4h
change in derived glucagon AUC | baseline (Day -1) to after dosing on Day 28
  change in pharmacodynamic parameters derived from glucagon; AUC0-4h

CONTACTS AND LOCATIONS:
Overall Officials: Yasuo Terauchi, MD, PhD, Principal Investigator — Yokohama City University
Locations (1):
- Yodogawaku, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/